CLINICAL TRIAL: NCT01927289
Title: A Double-blind Randomized Controlled Trial Between Ultrasound-guided Brachial Plexus and Distal Peripheral Nerve Blocks for Hand Surgery
Brief Title: DBRCT on the Effect of Grip Strength in Brachial Plexus vs Distal Forearm Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas Lam, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lamproxvsdistal
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Mobility
Keywords: Ultrasound; supraclavicular block; distal forearm block; Grip Strength; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proximal Brachial Plexus block (Active Comparator): 15 mls of 1.5% Mepivacaine injected in the supraclavicular approach and 15 mls of saline injected in the distal forarm nerve blocks
  Interventions: Procedure: Proximal Brachial Plexus vs Distal Forearm Block
- Distal Forearm block (Active Comparator): 15 mls 1.5% Mepivacaine injected in distal forearm nerve block and 15 mls of saline injected to the brachial plexus via the supraclavicular approach
  Interventions: Procedure: Proximal Brachial Plexus vs Distal Forearm Block

INTERVENTIONS:
Procedure: Proximal Brachial Plexus vs Distal Forearm Block — Proximal Brachial plexus block: 15 mls saline injected in distal forearm nerve block and 15 mls of 1.5% Mepivacaine injected to the brachial plexus via the supraclavicular approach.
  Distal forearm block: 15 mls 1.5% Mepivacaine injected in distal forearm nerve block and 15 mls of saline injected to the brachial plexus via the supraclavicular approach
  Other Names: Supracalvicular block; Wrist block

SUMMARY:
This is a double-blind prospective randomized control trial. The primary hypothesis is that the preservation of motor function is superior in distal forearm blocks compared to supraclavicular block. The secondary outcomes include patient satisfaction, surgeon's satisfaction, rate of block success, onset and duration of block.

ELIGIBILITY:
Inclusion criteria:

1. American Society of Anesthesiologists physical status I to III
2. Aged 18 and above
3. Able to provide own consent
4. Elective ambulatory surgery in the hand with an expected surgical time of less than 15 minutes that is normally performed with a peripheral nerve block covering the median and ulnar nerve distributions and intravenous sedation without general anesthesia

Exclusion criteria:

1) Surgery outside the median and ulnar nerve distribution in the hand 2) Bilateral surgery 3) body mass index of more than 45 kg/m2 (higher chance of failure) 4) neck or clavicle deformities 5) infection at the injection site 6) existing neurologic disease 7) insulin dependent diabetes 8) Diabetes with peripheral neuropathy or end organ damage 9) allergy to LA agents 10) coagulopathy 11) Past surgery on the same upper limb 12) Any other contraindication to supraclavicular block or forearm blocks 13) Contraindication to monitored anesthesia care with peripheral nerve block as the mode of anesthesia.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Grip Strength | 6 months
  Maximal Grip Strength x3 using dynanometer

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  Patient satisfaction on a linear numerical scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, MD, Principal Investigator — UNM
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States